CLINICAL TRIAL: NCT03295617
Title: Management of Giant Thoracic Disc Hernias by Thoracoscopy: Experience of 52 Cases
Acronym: GHTT
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/xx
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Giant Thoracic Herniation; Myelopathy
Keywords: spinal thoracic herniation; surgery; endoscopic approach; thoracic spine; minimal invasive access
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Thoracoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- spinal thoracic herniation
  Interventions: Procedure: Thoracoscopy

INTERVENTIONS:
Procedure: Thoracoscopy — Thoracoscopy surgery

SUMMARY:
Introduction: Giant thoracic disc herniation is a rare condition for which surgical treatment is indicated when there are signs of spinal cord injury. To date, several surgical techniques have been described in the treatment of this condition on small patient series. The main objective is to evaluate the long-term results of a series of 53 patients treated with a minimally invasive endoscopic procedure. The secondary objective is to explain our pre-operative planning and the technical details of our procedure. METHOD: Retrospective monocentric study on a cohort of patients treated in our department. The following medical data from our database are analyzed: Morbidity of operative gesture (duration of procedure, bleeding, postoperative complications), clinical results at the last follow-up visit (thoracic Japanese Orthopedic Association (JOA) score, Frankel score, parietal pain , ability to walk, wish to carry out the same intervention again if necessary). On the radiological level, we evaluated the quality of the resection (total, subtotal, incomplete and impossible), the reappearance of a border of cerebrospinal fluid perimedullary and the presence of an intramedullary T2 hyperintense signal MRI post- operative. All these data are collected and analyzed anonymously. Expected Results: We believe we can demonstrate that thoracoscopy is a valid therapeutic option in the treatment of thoracic disc herniation responsible for spinal cord compression. This with a low morbidity given the minimally invasive nature of the approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated on giant thoracic thoracic disc herniation between May 2001 and October 2016

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient operated on giant thoracic thoracic disc herniation between May 2001 and October 2016
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Japanese Orthopedic Association Score | 30 minutes

SECONDARY OUTCOMES:
Frankel score | 30 minutes
Parietal pain measured by visual analogic scale | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David Brauge, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France